CLINICAL TRIAL: NCT03759236
Title: Increasing Human Papillomavirus (HPV) Vaccine Uptake Via General Health Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 48789
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2020-02

CONDITIONS: Human Papilloma Virus
Keywords: Health Messaging; Health Education; Human Papilloma Virus; HPV Vaccination
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: Two clinics are randomized to receive the health messaging via SMS and the third clinic is randomized to receive standard CDC health education materials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Health Messaging via SMS (Experimental): Clinics randomized to this arm will receive the health messaging via SMS intervention. Flyers and information cards will be made available in all exam rooms and the waiting room, which contain information about the health messaging program. Patients must voluntarily elect to enroll in the program using their mobile device. Patients who enroll will receive a variety of health messages on topics including HPV Vaccine, Cervical Cancer screening, Birth Control options, Menstrual Problems, diet and exercise. Text messages are sent out using a third party interface, Twilio, at a frequency of 2 times each week for a duration of 1 year. These are one-way messages which only allow for texts to be sent to the participant.
  Interventions: Behavioral: Health Messaging via SMS
- CDC Pamphlets (Active Comparator): The clinic randomized to this control arm will receive standard Center for Disease Control health pamphlets about the HPV Vaccine. Flyers are posted in the clinic waiting room and exam room.
  Interventions: Behavioral: CDC Health Pamphlets

INTERVENTIONS:
Behavioral: Health Messaging via SMS — This intervention aims to provide health education on topics including HPV Vaccination, Cervical Cancer screening, contraceptive methods, menstrual problems, diet and exercise geared towards women with children of vaccination age.
  Arms: Health Messaging via SMS
Behavioral: CDC Health Pamphlets — This intervention aims to provide health education on the HPV Vaccination to women with children of vaccination age.
  Arms: CDC Pamphlets

SUMMARY:
Background: Prevention of cervical cancer and genital warts could be achieved by immunization with the prophylactic human papillomavirus (HPV) vaccines commercially available. However, in the U.S. only 38% of females and 14% of males in the recommended age group (9-26 years) receive the complete, three-dose HPV vaccine. Because the HPV vaccine is covered under the Vaccine for Children Program, the underinsured and uninsured have no-cost access. Nonetheless, data from Los Angeles county suggest that HPV vaccination rates among the uninsured and underinsured groups are significantly lower than the national average, likely related to knowledge of the vaccine, transportation, number of doses and concern of side effects.

Aim: To evaluate the efficacy of health oriented text messaging to increase HPV vaccine uptake versus standard health messaging (Center for Disease Control and Prevention (CDC) HPV vaccine information flyers).

Hypothesis: The investigators hypothesize that receiving general health messaging, including messages regarding the benefits of the HPV vaccine, will increase HPV vaccine uptake. Text messaging will also be more successful in reaching the uninsured and underinsured populations than will traditional flyers/information pamphlets used in clinics.

Methods: A cluster randomized trial design will be used to recruit participants from four clinics in Los Angeles County which offer pediatric vaccination to uninsured and underinsured children. The sample will include women aged 18-45 years of age. Two of the sites will be randomized to the text messaging arm and the other clinic will be randomized to the control arm (standard messaging: CDC flyers and pamphlets available for patients at the clinic). Outcome measures will be HPV vaccinations rates at those clinics. Rates will be defined into groups who received 1 dose, 2 doses and 3 doses.

Anticipated Results: The investigators expect to find statistically significant higher HPV vaccination rates among children and women in the text messaging study arm compared to the control arm.

Implications and Future Studies: This pilot study will give us preliminary data to submit a larger randomized controlled trial to examine the efficacy of text messaging.

DETAILED DESCRIPTION:
Prevention of cervical cancer and genital warts could be achieved by immunization with the prophylactic human papillomavirus (HPV) vaccines commercially available. However, in the U.S. only 38% of females and 14% of males in the recommended age group (9-26 years) receive the complete, three-dose HPV vaccine. Because the HPV vaccine is covered under the Vaccine for Children Program, the underinsured and uninsured have no-cost access. Nonetheless, data from Los Angeles county suggest that HPV vaccination rates among the uninsured and underinsured groups are significantly lower than the national average, likely related to knowledge of the vaccine, transportation, number of doses and concern of side effects. The primary objective of this pilot study is to evaluate the efficacy of health oriented text messaging to increase HPV vaccine uptake versus standard health messaging (Center for Disease Control and Prevention (CDC) HPV vaccine information flyers).

The investigators hypothesize HPV vaccine uptake will be improved through the receipt of general health messaging that includes HPV vaccine messages. Such messaging will increase knowledge about HPV vaccine availability, as well as improve the perceptions around HPV vaccination. Text messaging will also be more successful in reaching large population groups than traditional flyers/information pamphlets used in clinics.

First, among our three participating clinics, the investigators convened community advisory boards (CABs) of individuals who are English and Spanish speaking to identify appropriate text messages including content, length of message and frequency of messaging (once a week, every other week). Topics included HPV vaccine messages, contraceptive information on hormonal contraception, long-acting reversible contraceptive (LARC) methods, dysmenorrhea, frequent menses, and vaginal discharge. The investigators focused on all topics and specifically messaging of HPV vaccine that are considered neutral and yet compelling. The investigators built upon the feedback obtained from the CAB. Each clinic serves at least 500 uninsured and underinsured children that offer regular HPV vaccination to these children. Of these three clinics, two of the sites will be randomized to the intervention arm (text messaging) and 1 site to have CDC flyers only. The sites currently collect information on all immunization given at their site. The sites will de-identify their vaccine rates for HPV at the end of the study and send us the de-identified data sets for vaccine rates, age (not birth date) and number of nursing/doctor visits made by age group.

ELIGIBILITY:
Inclusion Criteria:

* Women who are patients at the clinic
* Age 21+
* Have a working mobile phone with SMS capability

Exclusion Criteria:

* Male
* <21 years of age
* Do not have a working mobile phone with SMS capability

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
HPV Vaccination Rate | 1 year
  In both arms of the study, we will collect data on the number of females aged 9- 26 years who made any visit to the clinic (denominator) and the number of females aged 9-26 vaccinated (numerator). Vaccination rates will be defined into groups who received at least 1 dose, compared to receiving none. We will also examine those receiving at least 2 doses vs 1 vs none.

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Barbara Moscicki, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No